CLINICAL TRIAL: NCT05624164
Title: Randomized Controlled Trial of Patients Treated With and Without Lateralized Microfracture During Rotator Cuff Repair
Brief Title: Microfracture at Proximal Humerus Lateral to Footprint Could Enhance the Rotator Cuff Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: micorfracture
Record Dates: First submitted 2022-10-30; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-08

CONDITIONS: Rotator Cuff Tears; Micro Fracture
Keywords: rotator cuff tear; microfracture
MeSH Terms: conditions — Rotator Cuff Injuries; Fractures, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateralized microfracture group (Experimental): Participants with medium to larger size rotator cuff tears will be treated with arthroscopy rotator cuff repair with microfracture at the lateral side of the footprint immediately.
  Interventions: Procedure: Lateralised microfracture
- No microfracture group (No Intervention): Participants with medium to larger size rotator cuff tears will be treated with arthroscopy rotator cuff repair without microfracture.

INTERVENTIONS:
Procedure: Lateralised microfracture — making microfracture(4 holes with 2mm diameter) at the lateral side of the footprint right after arthroscopy rotator repair.
  Arms: Lateralized microfracture group

SUMMARY:
The goal of this clinical trial is to test whether there is any effect on rotator cuff healing by making microfracture at the lateral side of the footprint. The main question it aims to answer are:

* [whether the lateralized microfracture could decrease the retear rate after arthroscopy rotator cuff repair.]
* [whether the lateralized microfracture could improve the functional recovery after arthroscopy rotator cuff repair.] Participants with medium to larger size rotator cuff tears will be randomly assigned to the study group treated with lateralized microfracture immediately after arthroscopy rotator cuff repair or the control group treated with conventional arthroscopy rotator cuff repair without microfracture.

ELIGIBILITY:
Inclusion Criteria:

1. Medium to large Rotator cuff tear(1cm-5cm) diagnosed by MRI
2. Patients can complete the follow-up and comply with all post-operative rehab instructions
3. Failure of non-operative treatment for at least 3 months

Exclusion Criteria:

1. Revision rotator cuff surgery
2. Partial thickness rotator cuff tears
3. Small (less than 1cm) and Massive (greater than 5cm) rotator cuff tears
4. Disease history of the affected shoulder
5. Systemic immune diseases
6. Irreparable rotator cuff tear

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | 24 months postoperative
  The scans were evaluated for rotator cuff integrity and degree of re-tears (no re-tears, partial or complete re-tear) by an independent radiologist

SECONDARY OUTCOMES:
Active range of motion of Shoulder | Preoperative, 3 months and 24 months postoperative
  Active forward flexion, abduction and external rotation will be measured with a manual goniometer at the preoperative visit, 3 months and 24 months after surgery.
Passive range of motion of Shoulder | Preoperative, 3 months and 24 months postoperative
  Passive forward flexion, abduction and external rotation will be measured with a manual goniometer at the preoperative visit, 3 months and 24 months after surgery.
American Shoulder and Elbow Score | Preoperative, 3 months and 24 months postoperative
  American Shoulder and Elbow scores (minimum 0 points, maximum 100 points, higher values are considered better outcomes) of patients with rotator cuff tears treated with and without lateralized microfracture at the preoperative visit, 3 months and 24 months after surgery.
University at California at Los Angeles Shouder Rating Scale | Preoperative, 3 months and 24 months postoperative
  University at California at Los Angeles Shoulder Rating Scale(minimum 3 points, maximum 35 points, higher values are considered better outcomes) of patients with rotator cuff tears treated with and without lateralized microfracture at the preoperative visit, 3 months and 24 months after surgery.
Visual Analog Scale for Pain | Preoperative, 3 months and 24 months postoperative
  Visual Analog Scale for Pain(minimum 0 points, maximum 10 points, higher values are considered worse outcomes) of patients with rotator cuff tears treated with and without lateralized microfracture at the preoperative visit, 3 months, and 24 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yucheng Sun, Ph.D, Principal Investigator — Affiliated Hospital of Nantong University
Locations (2):
- China (2):
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Afiliated Hospital of Nantong University, Nantong, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jo CH, Shin JS, Park IW, Kim H, Lee SY. Multiple channeling improves the structural integrity of rotator cuff repair. Am J Sports Med. 2013 Nov;41(11):2650-7. doi: 10.1177/0363546513499138. Epub 2013 Aug 13. PMID 23942284
- [Result] Orth P, Duffner J, Zurakowski D, Cucchiarini M, Madry H. Small-Diameter Awls Improve Articular Cartilage Repair After Microfracture Treatment in a Translational Animal Model. Am J Sports Med. 2016 Jan;44(1):209-19. doi: 10.1177/0363546515610507. Epub 2015 Nov 6. PMID 26546301
- [Result] de Girolamo L, Jannelli E, Fioruzzi A, Fontana A. Acetabular Chondral Lesions Associated With Femoroacetabular Impingement Treated by Autologous Matrix-Induced Chondrogenesis or Microfracture: A Comparative Study at 8-Year Follow-Up. Arthroscopy. 2018 Nov;34(11):3012-3023. doi: 10.1016/j.arthro.2018.05.035. Epub 2018 Sep 25. PMID 30266548
- [Result] Sun Y, Kwak JM, Kholinne E, Zhou Y, Tan J, Koh KH, Jeon IH. Small Subchondral Drill Holes Improve Marrow Stimulation of Rotator Cuff Repair in a Rabbit Model of Chronic Rotator Cuff Tear. Am J Sports Med. 2020 Mar;48(3):706-714. doi: 10.1177/0363546519896350. Epub 2020 Jan 13. PMID 31928410
- [Result] Steadman JR, Briggs KK, Rodrigo JJ, Kocher MS, Gill TJ, Rodkey WG. Outcomes of microfracture for traumatic chondral defects of the knee: average 11-year follow-up. Arthroscopy. 2003 May-Jun;19(5):477-84. doi: 10.1053/jars.2003.50112. PMID 12724676
- [Result] Osti L, Del Buono A, Maffulli N. Microfractures at the rotator cuff footprint: a randomised controlled study. Int Orthop. 2013 Nov;37(11):2165-71. doi: 10.1007/s00264-013-1952-z. Epub 2013 Jun 13. PMID 23760681
- [Result] Kida Y, Morihara T, Matsuda K, Kajikawa Y, Tachiiri H, Iwata Y, Sawamura K, Yoshida A, Oshima Y, Ikeda T, Fujiwara H, Kawata M, Kubo T. Bone marrow-derived cells from the footprint infiltrate into the repaired rotator cuff. J Shoulder Elbow Surg. 2013 Feb;22(2):197-205. doi: 10.1016/j.jse.2012.02.007. Epub 2012 Apr 28. PMID 22543003